CLINICAL TRIAL: NCT04576247
Title: Feasibility, Acceptability, and Effects of Combined Aerobic and Resistance Exercise in Breast Cancer Survivors: A Pilot Study (the CARE Study)
Brief Title: Combined Modality Exercise and Appetite in Breast Cancer Survivors
Acronym: CARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-3032.cc
Record Dates: First submitted 2020-09-15; First posted 2020-10-06 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer Female; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Masking Description: Masking is not possible because this is a single-arm exercise study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined aerobic and resistance exercise (Experimental): 12 weeks of supervised resistance exercise and unsupervised aerobic exercise.
  Interventions: Behavioral: Combined aerobic and resistance exercise

INTERVENTIONS:
Behavioral: Combined aerobic and resistance exercise — The 12-week intervention will build upon an ongoing resistance exercise program for cancer patients and survivors at the University of Colorado's Anschutz Health and Wellness Center. Resistance exercise will be led by certified cancer exercise specialists who provide individualized exercise programs to cancer patients and survivors. Exercise sessions are progressive, target all major muscle groups, are 50 minutes in duration, and completed 2x/week.
  The intervention will also include 3 self-directed moderate-intensity aerobic exercise sessions/week, building to 50 minutes at 60% heart rate maximum (determined at baseline). Target exercise will be achieved by a gradual progression of exercise duration over the first four weeks of the program.

SUMMARY:
The overall aim of this research is to assess the feasibility of a 12-week combined aerobic exercise (AEx) and resistance exercise (REx) intervention and elucidate the impact of AEx/REx on several physiological and behavioral components of energy balance among breast cancer survivors (BCS).

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age: 18 - 45 years
* Body mass index [BMI]: 25 - 35 kg/m2
* Pre-menopausal before cancer diagnosis and treatment
* <1 hour/week of planned physical activity by self-report in the previous 12 months
* Diagnosis of primary stage I - III estrogen receptor/progesterone receptor-positive (ER/PR+) breast cancer, according to institutional standards.
* All chemotherapy, radiation, and surgery completed at least two weeks (14 days), but less than 6 months prior to registration

Exclusion Criteria:

* Self-reported diabetes mellitus, untreated/uncontrolled thyroid disease, history of cardiovascular disease or symptoms suggestive of cardiovascular disease (chest pain, shortness of breath at rest or with mild exertion, syncope), cancer diagnosis in the last 5 years before breast cancer (any site, excluding skin cancer), or any other medical condition affecting weight or energy metabolism.
* Uncontrolled hypertension defined as: systolic blood pressure >160 mmHg or diastolic blood pressure >100mmHg, as measured during the screening visit. Participants who are deemed ineligible based upon uncontrolled hypertension criteria will be referred to their primary care physicians for treatment. If this condition becomes controlled they will be allowed to be re-evaluated for inclusion in the current trial.
* Unable to exercise due to cardiac, pulmonary, neurological, orthopedic reasons.
* Currently smoking and/or nicotine use.
* Treatment with medications known to significantly affect appetite, weight, energy intake or expenditure in the last 3 months (e.g. appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants).
* Corticosteroid use within the last two weeks
* History of surgical procedure for weight loss at any time (e.g. gastroplasty, gastric bypass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve); history of extensive bowel resection for other reasons
* Currently pregnant, lactating or less than 6 months post-partum.
* Score of ≥ 2 on the CAGE (cut-annoyed-guilty-eye opener) questionnaire adapted to include drug use55
* Score of > 20 on the Eating Attitude Test - 26 (EATS-26), indicative of disordered eating. Participants with a score >20 on the EATS-26 will be referred to their primary care physician for further evaluation.
* Significant food intolerances/allergies that cannot be accommodated by the University of Colorado Hospital Clinical Translational Research Center Metabolic Kitchen.
* Currently participating in any formal weight loss or physical activity programs or clinical trials for weight loss.
* Other medical, psychiatric, or behavioral limitations that may interfere with participation (as determined by study physician).
* Unable or unwilling to undergo study procedures

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Recruitment and enrollment feasibility | Through study completion, up to two years
  Number of individuals approached, meeting inclusion criteria, reasons for exclusion, and enrolled in the study
Subjective exercise adherence | Changes across weeks 4, 8, and 12
  Participants will be asked to rate on a 1-10 Likert scale: 1) how adherent they were to the prescribed exercise over the past week, 2) how difficult it was to adhere to the prescribed exercise over the past week, and 3) how likely they feel they can adhere to the prescribed exercise for the next month.
Exercise self efficacy | Changes across weeks 4, 8, and 12
  Self Efficacy for Exercise Scale; 9 items; score range: 0-9, with higher scores indicating higher exercise self-efficacy
Exercise enjoyment | Changes across weeks 4, 8, and 12
  Physical Activity Enjoyment Scale; 8 items; range: 7-56, with higher scores indicating higher exercise enjoyment
Intervention acceptability | 12 weeks
  Subjective ability to adhere to combined AEx/REx
Intervention acceptability | 12 weeks
  Barriers to completing AEx/REx
Intervention acceptability | 12 weeks
  Open-ended opinions on the structure and content of the exercise training sessions
Intervention acceptability | 12 weeks
  Changes in subjective physical function, cancer-specific side effects, and overall well-being directly related to the exercise intervention
Objective exercise adherence | 12 weeks
  Adherence to additional study-specific AEx will be tracked through heart rate monitor data, logs of attendance, and participant diaries and compared to the REx-only intervention

SECONDARY OUTCOMES:
Changes in ghrelin | Baseline, 12 weeks
  Fasting ghrelin, ghrelin area under the curve in response to a control meal
Changes in peptide-YY (PYY) | Baseline, 12 weeks
  Fasting PYY, PYY area under the curve in response to a control meal
Changes in subjective appetite ratings | Baseline, 12 weeks
  Changes in hunger, satiety, and prospective food consumption via visual analog scales
Changes in ad libitum energy intake | Baseline, 12 weeks
  Energy intake from buffet-style meal
Changes in physical activity | Baseline, 12 weeks
  Step count measured by accelerometers
Changes in sedentary behavior | Baseline, 12 weeks
  Time in sedentary activities measured by accelerometers

OTHER OUTCOMES:
Changes in resting energy expenditure | Baseline, 12 weeks
  Resting energy expenditure measured by metabolic cart and adjusted for body composition changes
Changes in body composition | Baseline, 12 weeks
  Fat mass and fat-free mass in kg, measured by dual X-ray absorptiometry
Changes in fatigue | Baseline, 12 weeks
  Measured by the Functional Assessment of Chronic Illness and Therapy - Fatigue; 13 questions; score range: 0-52, with higher score indicating higher fatigue

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Univeristy of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado Cancer Center, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No